CLINICAL TRIAL: NCT02536625
Title: RAPANK: Study of the Impact of Everolimus Treatment on the Development and Functions of Lymphocytes NK (Natural Killer), for Patients With a Metastatic Breast Cancer (HR+ / HER2/Neu Negative)
Brief Title: Study of the Impact of Everolimus Treatment on Lymphocytes NK (Natural Killer) Development and Functions for Patients With a Metastatic Breast Cancer (HR+ / HER2/Neu Negative)
Acronym: RAPANK
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Collaborators: The Biostatistics and Therapy Evaluation Unit (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: RAPANK
Record Dates: First submitted 2015-08-14; First posted 2015-09-01 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: everolimus; NK; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Prospective Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Everolimus: Immunomonitoring
  Interventions: Other: prospective study

INTERVENTIONS:
Other: prospective study

SUMMARY:
NK (Natural Killer) cells are important in the fight against tumor, especially for the control of cancer metastasis. The purpose of this prospective study is to evaluate the impact on lymphocytes NK functions and development of an everolimus treatment in women treated for a metastatic breast cancer. In particular, the study of lymphocytes NK functions and development under everolimus treatment could permit to validate an early biomarker of the impact of everolimus on these NK cells.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years old
* Metastatic breast cancer HR+ (Hormone Receptor positive), HER2/neu negative (Human Epidermal Growth Factor Receptor-2)
* ECOG PS (Eastern Cooperative Oncology Group Performance Status) ≤2
* Eligible to an hormonotherapy treatment combined to an mTOR (mammalian Target Of Rapamycin) inhibitor (i.e. SPC (Summary of Product Characteristics) modalities)
* Measurable disease according to RECIST 1.1 (Response Evaluation Criteria In Solid Tumors)
* Not receiving the non-authorized concomitant treatments
* Patient should understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed.
* Patients must be covered by a medical insurance

Exclusion Criteria:

* BMI>30
* All dysimmune disease, history of transplantation or immunosuppressive therapy or corticotherapy
* All chronic inflammatory diseases
* Last chemotherapy < 6 months
* Corticotherapy <1 year and more than 1 month
* Restrictive diet ≤3 months before inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With a Metastatic Breast Cancer (HR+ / HER2/Neu Negative) eligible for a treatment with everolimus in this application
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Measure of the level of Granzyme B (GzmB) | Timepoint at 3 months

SECONDARY OUTCOMES:
Objective Response Rate | 12 months
  The objective response rate (ORR) will be defined as the proportion of patients (described on the efficacy-evaluable population) who achieve complete response (CR) or partial response (PR). ORR is based on tumor assessments (measurements according to RECIST 1.1
Progression-Free Survival (PFS) | 12 months
  Measured from the date of study drugs start to the date of the first objective radiological disease progression using RECIST 1.1 or death.
Overall Survival (OS) | 12 months
  Defined as the duration of time from start of treatment to time of death.
Intercurrent diseases reporting | 12 months
  Number of patients with adverse events (including infectious events) related to everolimus
Circulating NK functions | Timepoint at 3 months and at 9 months
  Characterization of circulating NK functions by flow cytometry
mTOR activation status | Timepoint at 3 months and at 9 months
  rpS6 phosphorylation rate by western blot

CONTACTS AND LOCATIONS:
Overall Officials: TREDAN Olivier, MD, Principal Investigator — Centre Leon Berard
Locations (2):
- France (2):
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite